CLINICAL TRIAL: NCT03133494
Title: Comparing Arterial Blood Gas(ABG) in Laparoscopic Cholecystectomy Between Smokers and Non Smokers: A Randomized Double Blind Case Control Study
Brief Title: Arterial Blood Gas Analysis in Laparoscopic Cholecystectomy
Acronym: ABG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Banaras Hindu University (Other)
Responsible Party: Principal Investigator, Amiya Kumar Barik, abarik, Final year resident, Department of Anesthesiology, Institute of Medical Sciences, Banaras Hindu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 2014-15/EC/1219
Record Dates: First submitted 2017-03-12; First posted 2017-04-28 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Cholecystectomy, Laparoscopic

STUDY DESIGN:
Intervention Model Description: Arterial blood gas sample was drawn from both the groups and analysed for any change in the desired parameters
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic cholecystectomy in smokers (Active Comparator): ABG analysis of patients with history of smoking posted for laparoscopic cholecystectomy was collected
  Interventions: Other: ABG analysis
- Laparoscopic cholecystectomy nonsmokers (Placebo Comparator): ABG analysis of patients without history of smoking posted for laparoscopic cholecystectomy was collected
  Interventions: Other: ABG analysis

INTERVENTIONS:
Other: ABG analysis — ABG analysis was performed and compared between two groups

SUMMARY:
The investigator found out that as such the base line carbon dioxide (CO2) level is higher in smokers as compared to non-smokers even before creation of pneumoperitoneum, which is due to the compromised lung function following chronic smoking. This condition gets aggravated after creation of pneumoperitoneum which is very much evident from the serial arterial blood gas analysis. The level of CO2 remains elevated even after deflation of the pneumoperitoneum. Hence one has to be very much vigilant not only during intra-operative period but also in post-operative care unit. Hence serial ABG monitoring should be included as a part of the protocol especially in laparoscopic surgeries.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy procedure is the treatment of choice for cholelithiasis as it has several advantages like smaller and more cosmetic incision, reduced blood loss, less postoperative pain, reduced post-operative stay, low post-operative complications, and early mobilization. Although this type of surgery is minimally invasive in nature but creation of pneumoperitoneum and postural changes causes a number of physiological alterations. Carbon dioxide (CO2) is the most commonly used gas for this purpose because it does not support combustion, is cleared more rapidly than other gases, and is highly soluble in blood. However, the disadvantage of CO2 is that the absorption of CO2 can cause hypercapnia and respiratory acidosis. Hypercapnia activates the sympathetic nervous system leading to an increase in blood pressure, heart rate, arrhythmias and myocardial contractility as well as it also sensitizes myocardium to catecholamines. Increased IAP may compress venous vessels causing an initial increase in preload, followed by a sustained decrease in preload.

Tobacco smoking is an internationally accepted health hazard. The United nation (UN) health agency reports that about 4.9 million people die each year across the globe due to cigarette smoking. Chronic smoking (more than 20 pack year at least for 10 year) causes a number of pathological changes in respiratory system which includes inflammatory changes in lung parenchyma, imbalance between protease and anti-protease, oxidative stress, cilliary dysfunction, mucosal hyper secretion, airflow limitation and pulmonary hypertension.

Arterial blood gas analysis plays a very important role in assessing the acid-base status, adequacy of oxygenation and ventilation. It is very useful in management of critically ill patients and in patients with pulmonary disorders. It is also a standard part of work-up for the patients who present with unexplained hypoxemia and dyspnea. An ABG test uses blood drawn from an artery, where the oxygen and carbon dioxide levels can be measured before they enter body tissues.

ELIGIBILITY:
Inclusion Criteria:

* American society of Anesthesiology (ASA) grade 1 and 2
* History of smoking (more than 20 pack year) for more than 10years

Exclusion Criteria:

* Patients refusal
* ASA grade 3 and 4
* Other lung pathologies
* Other cardiac pathologies
* uncontrolled diabetes mellitus
* systemic infection
* emergency operation
* history of malignancy
* history of alcohol or drug abuse

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2016-04-01 (Actual); Study Completion 2016-04-01 (Actual)

PRIMARY OUTCOMES:
Arterial blood gas parameter like potential of hydrogen (PH) | 10 minutes before starting to 30 minutes after completion of surgery
  Above parameter was measured by serial ABG analysis

SECONDARY OUTCOMES:
Arterial blood gas parameter like partial pressure of carbon dioxide (PCO2) | 10 minutes before starting to 30 minutes after completion of surgery
  Above parameter was measured by serial ABG analysis
Arterial blood gas parameter like bicarbonate(HCO3) | 10 minutes before starting to 30 minutes after completion of surgery
  Above parameter was measured by serial ABG analysis
Arterial blood gas parameter like base excess (BE) | 10 minutes before starting to 30 minutes after completion of surgery
  Above parameter was measured by serial ABG analysis

CONTACTS AND LOCATIONS:
Overall Officials: PUSKAR RANJAN, MD, PhD, Principal Investigator — Banaras Hindu University

IPD SHARING:
Plan to Share IPD: Undecided